CLINICAL TRIAL: NCT03442283
Title: Supplemental Vitamins and Minerals for CVD Prevention and Treatment: Systematic Review and Meta-analyses of the Data (Meta-analyses and RCTs) Published Since 2012
Brief Title: Meta-analysis of Randomized Controlled Trials on Vitamins and Mineral Supplementation for CVD Prevention and Treatment
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, David Jenkins, Professor, University of Toronto
Other Study IDs: META SUPPLEMENTS 001
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Cardiovascular Diseases
Keywords: Supplements, Cardiovascular Diseases, All-cause mortality, Meta-Analysis
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Supplementation
  Interventions: Dietary Supplement: Vitamin mineral supplementation
- No Supplementation

INTERVENTIONS:
Dietary Supplement: Vitamin mineral supplementation — supplementation with a vitamin or mineral: vitamin A, β-carotene, B1, B2, B3 (niacin), B6, B10 (folic acid), C, D and E, calcium, iron, zinc, magnesium and selenium. Also, multivitamins, antioxidants, B-complex and the combination of calcium and vitamin D.
  Groups: Supplementation

SUMMARY:
The use of vitamin and mineral supplementation has historically been to treat and prevent micronutrient deficiencies. In recent years, however, and with their widespread use, the interest has shifted toward a possible role in the prevention and treatment of chronic diseases. The investigators will review and perform meta-analyses of vitamin and mineral supplementation trials in relation to cardiovascular disease. Publications from 2012, both before and including the US Preventive Service Task Force (USPSTF) 2014 review, will be included in the review.

DETAILED DESCRIPTION:
Search strategy:

A literature search of the Cochrane Library, Medline and PubMed will be conducted with the following search terms: "dietary supplements or supplement*" AND "cardiovascular disease or myocardial infarction or stroke or cardiovascular death or mortality or all-cause mortality or death." Specific searches will be conducted for individual supplements and included multivitamins, antioxidants, vitamin A, β-carotene, B1, B2, B3 (niacin), B6, B10 (folic acid), B-complex, C, D and E, calcium, iron, zinc, magnesium and selenium. The search will be limited to meta-analyses and RCTs.

Analysis:

Full article review and data extraction will be conducted by two independent investigators, with all disparities reconciled through consensus. The extracted data will include number of cases and total participants/population for the intervention and control group.

Data will be analyzed using Review Manager (RevMan) version 5.3 (The Nordic Cochrane Centre, The Cochrane Collaboration, Copenhagen, Denmark) and publication bias will be conducted using STATA software, version 13.0 (College Station, TX, USA). Heterogeneity will be assessed using the Cochran Q statistic at p<0.1 and quantified by the I² statistic. Publication bias will be investigated by visual inspection of funnel plots and quantitative assessment using Begg's and Egger's tests where p<0.05 is considered evidence of small study effects. If <10 trials are available in a meta-analysis, publication bias analysis will not be assessed due to insufficient power.

Risk of bias The Cochrane risk of bias tool which is based on randomization, allocation concealment, blinding, completeness of follow-up and intention-to-treat will be used to assess eligible RCTs.

Grading of the evidence The quality and strength of the evidence will be assessed using the Grading of Recommendations Assessment, Development, and Evaluation (GRADE) tool. Using the GRADE tool, evidence will be graded as high, moderate, low, or very low quality evidence using the following criteria: study limitations (as assessed by the Cochrane Risk of Bias Tool), inconsistency (substantial) unexplained inter-study heterogeneity, I2>50% and p<0.1; indirectness (presence of factors that limit the generalizability of the results); imprecision (the 95% CI for effect estimates crosses a minimally important difference (MID) of 5% [RR 0.95-1.05]) from the line of unity; and publication bias (significant evidence of small-study effects).

ELIGIBILITY:
Inclusion Criteria:

* English studies
* Supplements taken orally for at least 6 months

Exclusion Criteria:

* Studies in children
* Studies in women who are pregnant or breastfeeding
* Studies of adults who have serious chronic disease infections such as HIV
* Studies with combined interventions and no adequate control group (i.e. interventions other than the supplement must be provided to the control group as well)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults free of serious chronic disease infections.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular disease (CVD) | 1 year
Coronary heart disease (CHD) | 1 year
Myocardial infarction (MI) | 1 year
Stroke | 1 year
CVD mortality | 1 year
CHD mortality | 1 year
MI mortality | 1 year
stroke mortality | 1 year
All-cause mortality | 1 year

IPD SHARING:
Plan to Share IPD: No